CLINICAL TRIAL: NCT00842270
Title: A Multicenter, Double-blind, Placebo-controlled, Randomized, Parallel-group Study to Evaluate the Efficacy of Oral AB1010 in Adult Patients With Severe Persistent Corticosteroid Dependent Asthma
Brief Title: Efficacy of Oral AB1010 in Adult Patients With Severe Persistent Corticosteroid Dependent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AB Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB04026
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Asthma
Keywords: severe asthma; corticosteroids dependent; asthma exacerbation; weaning; tyrosine kinase inhibitor; severe persistent corticosteroid dependent asthma
MeSH Terms: conditions — Asthma | interventions — masitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2 (Experimental): 4,5 mg/kg/day
  Interventions: Drug: AB1010
- 3 (Experimental): 6 mg/kg/day
  Interventions: Drug: AB1010
- 4 (Placebo Comparator): matching placebo for AB1010 3, 4,5 and 6 mg/kg/day
  Interventions: Drug: placebo
- 1 (Experimental): AB1010 3 mg/kg/day
  Interventions: Drug: AB1010

INTERVENTIONS:
Drug: AB1010 — 3 mg/kg/day
  Other Names: masitinib
  Arms: 1
Drug: AB1010 — 4,5 mg/kg/day
  Other Names: masitinib
  Arms: 2
Drug: AB1010 — 6 mg/kg/day
  Other Names: masitinib
  Arms: 3
Drug: placebo — matching placebo to AB1010 dosages
  Arms: 4

SUMMARY:
The aim of the study is to evaluate, comparatively to a placebo, the activity of oral AB1010, administered at three dose levels during 4 months to patients with severe persistent corticosteroid dependent asthma, assessed on :

* the decrease in corticosteroid therapy
* the asthma control improvement (symptomatic scores, rescue medication intake, respiratory function)
* the pharmacokinetic profile of AB1010
* clinical and biological safety parameters

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, parallel-groups, multicenter study of daily oral AB1010 at doses 3, 4.5 and 6 mg/kg/day.

The study treatment is administered for 16 weeks:

* the first 4 weeks are a run-in period during which corticosteroids remain stable;
* during the following 8 weeks, corticosteroids are decreased every week until weaning or an exacerbation occurs;
* the last 4 weeks are a stabilization period. Patients have to perform a visit every 2 weeks during run-in, then every week for the following 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Known severe persistent corticosteroid dependent asthma (WHO/NHLBI workshop definition).
* Disease duration > 1 year.
* Stable disease with no exacerbation episode for at least one month before inclusion.
* Daily treated with 10 to 50 mg of equivalent prednisolone, with stable dosage since at least 3 months.
* Known reversibility of bronchial obstruction, defined as an enhancement of FEV1 ≥ 12%, 10 minutes after salbutamol administration, or 14 days after systemic treatment with 1 mg/kg/day of equivalent prednisolone.

Exclusion Criteria:

* Asthmatic patients still exposed to allergens or to triggering factors influencing asthma control.
* History of infection requiring hospitalization or treatment with antibiotics within 2 weeks of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-01; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
decrease in oral corticosteroid therapy (weaning extent) | 16 weeks

SECONDARY OUTCOMES:
asthma control improvement | 16 weeks
asthma exacerbation rate | 16 weeks

REFERENCES:
- [Background] Lee-Fowler TM, Guntur V, Dodam J, Cohn LA, DeClue AE, Reinero CR. The tyrosine kinase inhibitor masitinib blunts airway inflammation and improves associated lung mechanics in a feline model of chronic allergic asthma. Int Arch Allergy Immunol. 2012;158(4):369-74. doi: 10.1159/000335122. Epub 2012 Apr 4. PMID 22487554
- [Result] Humbert M, de Blay F, Garcia G, Prud'homme A, Leroyer C, Magnan A, Tunon-de-Lara JM, Pison C, Aubier M, Charpin D, Vachier I, Purohit A, Gineste P, Bader T, Moussy A, Hermine O, Chanez P. Masitinib, a c-kit/PDGF receptor tyrosine kinase inhibitor, improves disease control in severe corticosteroid-dependent asthmatics. Allergy. 2009 Aug;64(8):1194-201. doi: 10.1111/j.1398-9995.2009.02122.x. PMID 19614621